CLINICAL TRIAL: NCT03067285
Title: A Phase IV, Open-label, Randomised, Pilot Clinical Trial Designed to Evaluate the Potential Neurotoxicity of Dolutegravir/Lamivudine/Abacavir in Neurosymptomatic HIV Patients and Its Reversibility After Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide. DREAM Study
Acronym: DREAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA 9016
Record Dates: First submitted 2017-02-14; First posted 2017-03-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A phase IV, open-label, randomised, pilot clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Patients who postpone switching from DTG/3TC/ABC to ELV/COBI/FTC/TAF four weeks:
  Interventions: Drug: DTG/3TC/ABC + ELV/COBI/FTC/TAF
- Arm 2 (Experimental): Patients who switch from DTG/3TC/ABC to ELV/COBI/FTC/TAF during the baseline visit
  Interventions: Drug: ELV/COBI/FTC/TAF

INTERVENTIONS:
Drug: ELV/COBI/FTC/TAF — Treatment with ELV/COBI/FTC/TAF during 24 weeks since randomized.
  Arms: Arm 2
Drug: DTG/3TC/ABC + ELV/COBI/FTC/TAF — Patients continuing on treatment with DTG/3TC/ABC after the randomization for 4 weeks, and then switch to ELV/COBI/FTC/TAF for 24 weeks
  Arms: Arm 1

SUMMARY:
A phase IV, multicentre, randomised, open-label, pilot clinical trial designed to evaluate HIV-infected, aviremic patients who receive treatment with the combination of DTG/3TC/ABC and who have neuropsychiatric adverse effects that, in the opinion of the investigators, may be related to taking DTG/3TC/ABC, if they improve after switching antiretroviral therapy to the combination of ELV/COBI/FTC/TAF.

DETAILED DESCRIPTION:
we estimate that 64 participants will need to be enrolled in the study to demonstrate symptomatic improvement after switching antiretroviral therapy from DTG/3TC/ABC to ELV/COBI/FTC/TAF.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years of age diagnosed with HIV using normal serology techniques.
* Current antiretroviral therapy with DTG/3TC/ABC.
* HIV viral load < 50 copies/mL for at least 12 weeks prior to signing the consent form [(]confirmed by two assays at least 12 weeks apart with viremia < 50 copies/mL between both). If the patient has a recent routine blood test available (≤ 4 weeks) that includes determining HIV viral load, these results may be used for the screening visit. If this test is not available, or the test is more than four weeks old, viral load will be determined on the day of screening in order to confirm that the patient meets this criterion.
* Appearance or worsening of the following symptoms compared to when DTG/3TC/ABC was started:

  * Symptoms of anxiety or depression
  * Insomnia or other sleep disturbances
  * Headache
  * Cognitive complaints (attention, concentration or memory)
  * Alterations in behaviour (irritability, aggressiveness or agitation)
  * Dizziness of neurological or neurologically-mediated origin

Exclusion Criteria:

* Determination of at least one HIV viral load ≥ 50 copies/mL in the last 12 weeks.
* Allergy, intolerance or existence of resistance mutations to any of the components of ELV/COBI/FTC/TAF
* History of active CNS infections
* Active psychosis, major depression with psychotic symptoms or autolytic ideation
* Dementia or mental retardation
* Drug use with a diagnosis of abuse or dependence according to DSM-5 criteria
* Illnesses that may interfere with the study procedures
* Claustrophobia
* Presence of magnetisable devices in the body
* Inability to complete any of the study procedures
* Pregnant or nursing women, as well as women of childbearing age who do not agree to use an adequate birth control method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
To compare changes in the severity of neuropsychiatric symptoms potentially associated with the use of DTG/3TC/ABC, perceived by patients randomised to begin isolated symptomatic treatment or treatment associated with switching antiretroviral therapy. | Week 4
  To compare, between the two arms of the study, changes in the percentage and in the severity of neuropsychiatric symptoms compiled using the ACTG adverse effects scale.
  anxiety and depression scale.
To compare changes in the severity of neuropsychiatric symptoms potentially associated with the use of DTG/3TC/ABC, perceived by patients randomised to begin isolated symptomatic treatment or treatment associated with switching antiretroviral therapy. | Week 4
  To compare, between the two arms of the study, changes in the percentage and in the severity of neuropsychiatric symptoms compiled using the pittsburgh sleep quality index.
To compare changes in the severity of neuropsychiatric symptoms potentially associated with the use of DTG/3TC/ABC, perceived by patients randomised to begin isolated symptomatic treatment or treatment associated with switching antiretroviral therapy. | Week 4
  To compare, between the two arms of the study, changes in the percentage and in the severity of neuropsychiatric symptoms compiled using the depression scale.

SECONDARY OUTCOMES:
To evaluate changes in the severity of neuropsychiatric symptoms potentially associated with the use of DTG/3TC/ABC after switching to ELV/COBI/FTC/TAF | Week 4
  To evaluate the change in the percentage and in the severity of neuropsychiatric symptoms compiled using the ACTG adverse effects scale.
To evaluate changes in the severity of neuropsychiatric symptoms potentially associated with the use of DTG/3TC/ABC after switching to ELV/COBI/FTC/TAF | Week 4
  To evaluate the change in the percentage and in the severity of neuropsychiatric symptoms compiled using the pittsburgh sleep quality index
To evaluate changes in the severity of neuropsychiatric symptoms potentially associated with the use of DTG/3TC/ABC after switching to ELV/COBI/FTC/TAF | Week 4
  To evaluate the change in the percentage and in the severity of neuropsychiatric symptoms compiled using the hospital anxiety and depression scale.
To evaluate changes in neurocognitive function and volumetric, spectroscopic, tractographic and cerebral perfusion markers, acquired by Magnetic Resonance Imaging, after switching from DTG/3TC/ABC to ELV/COBI/FTC/TAF | Week 24 after the switching
  To evaluate the change in global neurocognitive function (global deficit score) and cognitive domains (T-scores) in the volumes of the different structures of the brain using MRI volumetric techniques; the change in levels of neuronal integrity estimated by determining N-acetylaspartate levels in the structures of the frontal lobe and the basal ganglia using spectroscopy.
To evaluate changes in neurocognitive function and volumetric, spectroscopic, tractographic and cerebral perfusion markers, acquired by Magnetic Resonance Imaging, after switching from DTG/3TC/ABC to ELV/COBI/FTC/TAF | Week 24 after the switching
  To evaluate the change in global neurocognitive function (global deficit score) and cognitive domains (T-scores) in the volumes of the different structures of the brain using MRI volumetric techniques; the change in the levels of white matter integrity estimated using the diffusion tensor imaging MRI technique.
To evaluate changes in neurocognitive function and volumetric, spectroscopic, tractographic and cerebral perfusion markers, acquired by Magnetic Resonance Imaging, after switching from DTG/3TC/ABC to ELV/COBI/FTC/TAF | Week 24 after the switching
  To evaluate the change in global neurocognitive function (global deficit score) and cognitive domains (T-scores) in the volumes of the different structures of the brain using MRI volumetric techniques; the change in the levels of brain inflammation estimated by determining the levels of choline and myo-inositol in the structures of the frontal lobe and basal ganglia using spectroscopy.
Percentages of virologic failure | Week 24 after the switching
  To evaluate the percentages of virologic failure after switching antiretroviral therapy from DTG/3TC/ABC to ELV/COBI/FTC/TAF

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Univ. Infanta Leonor, Madrid
  - Hospital Univ. La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No